CLINICAL TRIAL: NCT01019564
Title: Complete Easy Rub Comparative Efficacy Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: COMP-319-9424
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Myopia; Hyperopia; Astigmatism
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Easy Rub MPS (Experimental): Complete Easy Rub Formula MPS
  Interventions: Device: Complete Easy Rub Formula MPS
- Aquify MPS (Active Comparator)
  Interventions: Device: Aquify MPS

INTERVENTIONS:
Device: Complete Easy Rub Formula MPS — Multi-purpose solution
  Arms: Easy Rub MPS
Device: Aquify MPS — Multi-purpose solution
  Arms: Aquify MPS

SUMMARY:
The aim of this trial is to assess Complete Easy Rub compared to a competitor multi-purpose solution in terms of lens cleanliness, subjective response and ocular response, when lenses are worn bilaterally on a daily wear basis for two months.

The hypotheses for this trial are:

* Lens cleanliness measures between solutions will be no different.
* Subjective ratings between solutions will be no different.
* Ocular response between solutions will be no different.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and comprehend English and give informed consent as demonstrated by signing a record of informed consent;
* Be at least 18 years old, male or female;
* Willing to comply with the wearing and clinical trial visit schedule as directed by the investigator;
* Have ocular health findings considered to be "normal" and which would not prevent the participant from safely wearing contact lenses;
* Is correctable to at least 6/12 (20/40) or better in each eye with contact lenses;
* Able to successfully wear one of the lens types to be used in this study on a daily wear (DW) basis in conjunction with any multi-purpose contact lens care solution (not including hydrogen peroxide-based systems) for at least one month prior to allocation of test or control solution;

Exclusion Criteria:

* Any pre-existing ocular irritation, injury or condition (including keratoconus and herpes keratitis) of the cornea, conjunctiva or eyelids that would preclude contact lens fitting and safe wearing of contact lenses;
* Any systemic disease that adversely affects ocular health e.g. diabetes, Graves disease, and auto-immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjögrens syndrome and systemic lupus erythematosus. Conditions such as systemic hypertension and arthritis do not automatically exclude prospective participants;
* Use of, or a need for, concurrent category S3 and above ocular medication at enrolment and/or during the study;
* Use of, or a need for, any systemic medication or topical medications which may alter normal ocular findings/are known to affect a participant's ocular health/physiology or contact lens performance either in an adverse manner or beneficial manner at enrolment and/or during the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of lens cleanliness of test and control solutions when used with soft lenses at the end of the manufacturer-recommended replacement interval. | Day 30